CLINICAL TRIAL: NCT02900495
Title: Transcutaneous Electric Nerve Stimulation (TENS) for the Treatment of Nocturnal Enuresis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other); Albany Medical College (Other)
Responsible Party: Principal Investigator, Adam S Howe, Assistant Professor of Surgery, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS16-0389
Record Dates: First submitted 2016-08-28; First posted 2016-09-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Nocturnal Enuresis; Bedwetting
Keywords: Nocturnal Enuresis; Bedwetting; TENS
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Suprapubic TENS (Experimental): electrodes, 'transcutaneous electric nerve stimulation' placed onto the lower abdomen in the suprapubic region directly over the bladder
  Interventions: Device: transcutaneous electric nerve stimulation
- Posterior Tibial TENS (Experimental): electrodes, 'transcutaneous electric nerve stimulation' placed over the posterior tibial nerve behind the medial malleolus of the ankle and another electrode on the bottom of the foot
  Interventions: Device: transcutaneous electric nerve stimulation
- Parasacral TENS (Experimental): electrodes, 'transcutaneous electric nerve stimulation' placed over the S3 foramen on the sacrum on each side of the midline in the lower back/upper buttocks
  Interventions: Device: transcutaneous electric nerve stimulation
- Shoulder TENS (Placebo Comparator): electrodes, 'transcutaneous electric nerve stimulation' placed over the scapula on the shoulder/back
  Interventions: Device: transcutaneous electric nerve stimulation

INTERVENTIONS:
Device: transcutaneous electric nerve stimulation — electrodes placed per treatment arm, performed at bedtime, session time 15 min, frequency setting of 10 Hz, intensity setting to patient's tolerance, duration 30 days
  Other Names: TENS unit

SUMMARY:
Children referred to the pediatric urology clinic for primary nocturnal enuresis will be screened for enrollment. Patients who fail behavioral therapy and who meet inclusion criteria will be offered therapy with a TENS unit.

Patients will be randomized into four groups. Group 1 will be the direct bladder stimulation arm with electrodes placed onto the abdomen in the suprapubic region directly over the bladder. Group 2 will be the distal neural loop arm with electrodes placed over the posterior tibial nerve. Group 3 will be the proximal neural loop arm with electrodes placed about 2-3 cm lateral to the midline in the sacral region at the level of S3. Group 4 will be the control arm with electrodes placed on the scapula. We will aim to recruit 32 patients per group for a total of 128 patients. The patients will be provided with a TENS unit (TENS 3000 Analog) and electrode pads and caretakers instructed on how to use the apparatus.

The TENS sessions will be performed nightly before bed for 15 minutes. TENS units will be set at a frequency of 10 Hz, and intensity determined by the sensitivity threshold of the patient. Diaries including nighttime incontinence episodes and a "wet sheet" scale (dry, damp, wet, soaked) will be recorded, along with any adverse reactions to the TENS unit. Patients will be followed up after one month of TENS with evaluation including the Pediatric Urinary Incontinence Questionnaire, a validated tool for measuring quality of life in children with bladder dysfunction; this questionnaire will be filled out prior to starting TENS treatment in order to compare the effect of treatment on QOL. . They will then follow up on these parameters again after another month (one month off of TENS therapy) to assess the durability of treatment effect. The data will be collected at different time points (baseline, 1 month, 2 months) for each group by itself and the groups compared against each other using statistical analysis.

DETAILED DESCRIPTION:
Institutional review board was obtained. Children ages 5-18 years old referred to the pediatric urology clinic for primary nocturnal enuresis will be screened for enrollment. Behavioral therapy (limiting evening drinking, double voiding prior to bedtime, bowel habits, social anxiety factors) will be utilized first. Patients who fail will next be offered therapy with a bedwetting alarm device or a TENS unit as an alternative, and those who chose TENS therapy will be included in the study. Patients who have previously tried pharmacologic treatment for nocturnal enuresis, neuromodulation or other alternative therapy for urologic disorders, daytime incontinence symptoms, known "high volume" voiders (determined from history), bedwetting episodes on the average of less than two times per week, medications predisposing to incontinence (eg, Lithium for bipolar disorder), other known voiding or neurologic disorders (eg, overactive bladder, myelomeningocele), secondary etiologies for nocturnal enuresis (eg, cystitis, obstructive sleep apnea, urinary fistulae), and any contraindications to usage of a TENS unit such as having a pacemaker will be excluded. Patients who have previously tried the bedwetting alarm will not be excluded from the study. 128 patients will be chosen for enrollment into the study.

The patients will be randomized into four groups of 32 patients each. Group 1 will be the direct bladder stimulation arm with electrodes placed onto the abdomen in the suprapubic region directly over the bladder. Group 2 will be the distal neural loop arm with electrodes placed onto the bottom of the feet. Group 3 will be the proximal neural loop arm with electrodes placed about 2-3 cm lateral to the midline in the sacral region at the level of S3. Group 4 will be the sham arm with electrodes placed on the scapula. We will aim to recruit 32 patients per group for a total of 128 patients. Detailed explanation of the purpose of the study, along with the risks and benefits of TENS will be given to the patient and caretakers by a provider prior to obtaining informed consent for enrollment into the study. The patients will be provided with a TENS unit and electrode pads and caretakers instructed on how to use the apparatus.

Parents of enrolled patients will fill out nightly voiding diaries, recording nighttime incontinence episodes and subjective "wet sheets" scale per night (dry, damp, wet, soaked) for 30 days prior to randomization into the treatment arms. The TENS sessions will be performed nightly at bedtime for 15 minutes for 30 days. TENS units will be set at a frequency of 10 Hz, and intensity determined in the office by the sensitivity threshold of the patient. Voiding diaries will be kept each night while on TENS therapy, additionally recording which TENS setting was used, duration of therapy each night, and any adverse reactions to the TENS unit or increased symptoms (these patients will be terminated from the study and included as a treatment failure). Diaries will then be kept for 30 days after TENS therapy was completed to assess durability of treatment effects. At voiding diary day 30 (before first TENS treatment), day 60 (after completion of TENS therapy), and day 90 (one month off of TENS), patients and families will fill out the Pediatric Urinary Incontinence Questionnaire (PIN-Q), a validated tool for measuring quality of life in children with bladder dysfunction. Patients will follow up at days 0, 30, 60, 90, and as needed (worsening symptoms, adverse reactions, concerns, and questions regarding usage of TENS). Parents will be called on a weekly basis throughout the study to ensure compliance and address any questions or concerns. The results of mean nightly incontinence episodes, mean "wet sheets" scale score (0-3), and PIN-Q will be measured between time points (baseline, 1 month, 2 months for each group by itself and the groups compared against each other using statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* primary nocturnal enuresis
* wet nights occur more than once per week on average
* Failed Behavioral therapy treatment (limiting evening drinking, double voiding prior to bedtime, bowel habits, social anxiety factors)
* ability to provide informed consent and complete study requirements

Exclusion Criteria:

* the use of medications for nocturnal enuresis (DDAVP, imipramine, anticholinergics) less than 30 days from time of appointment
* daytime incontinence
* Known "high volume" voiders
* medications predisposing to incontinence (eg, Lithium for bipolar disorder)
* other known voiding or neurologic disorders (eg, overactive bladder, spina bifida, interstitial cystitis)
* secondary etiologies for nocturnal enuresis (cystitis, obstructive sleep apnea, urinary fistula)
* any contraindication to TENS unit usage (pacemaker or other implantable devices, lymphedema, pregnancy, malignancy)
* Any history of heart disease or complications

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Wet nights | 60 days
  Total number of change in wet nights compared in each TENS arm to control and baseline wet nights

SECONDARY OUTCOMES:
Severity | 60 days
  compare monthly mean "wet scale" score of each TENS arm to control and baseline score
Patient compliance | 60 days
  assess patient tolerance to TENS therapy and ability to perform TENS therapy at home (correct session time, settings, and consistency of use)
Quality of Life Scores | 60 days
  compare PIN-Q scores at initial visit, after baseline month, after one month of using TENS
Adverse reactions | 60 days
  record any adverse reactions to TENS therapy
Durability | 90 days
  compare patient response, monthly number of wet nights, "wet scale" score (severity), and PIN-Q score (quality of life) of each TENS arm one month after stopping TENS and compare to baseline data and immediately after one month of TENS therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lane S Palmer, MD, Principal Investigator — Cohen Children's Medical Center of NY
Locations (5):
- United States (5):
  - Albany Medical College, Albany, New York
  - Pediatric Urology Associates, Brooklyn, New York
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Pediatric Urology Associates, New Hyde Park, New York
  - Pediatric Urology Associates, Tarrytown, New York

IPD SHARING:
Plan to Share IPD: No
No plans to share this information

REFERENCES:
- [Result] Kajbafzadeh AM, Sharifi-Rad L, Mozafarpour S, Ladi-Seyedian SS. Efficacy of transcutaneous interferential electrical stimulation in treatment of children with primary nocturnal enuresis: a randomized clinical trial. Pediatr Nephrol. 2015 Jul;30(7):1139-45. doi: 10.1007/s00467-014-3039-5. Epub 2015 Jan 25. PMID 25618771
- [Result] Lordelo P, Benevides I, Kerner EG, Teles A, Lordelo M, Barroso U Jr. Treatment of non-monosymptomatic nocturnal enuresis by transcutaneous parasacral electrical nerve stimulation. J Pediatr Urol. 2010 Oct;6(5):486-9. doi: 10.1016/j.jpurol.2009.11.005. PMID 20837326
- [Result] Barroso U Jr, Lordelo P, Lopes AA, Andrade J, Macedo A Jr, Ortiz V. Nonpharmacological treatment of lower urinary tract dysfunction using biofeedback and transcutaneous electrical stimulation: a pilot study. BJU Int. 2006 Jul;98(1):166-71. doi: 10.1111/j.1464-410X.2006.06264.x. PMID 16831163
- See also: Pediatric Urology Associates, P.C. — http://www.pedsurology.com/

DOCUMENTS (1):
  • Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT02900495/ICF_000.pdf